CLINICAL TRIAL: NCT07246668
Title: A Phase II Single-Arm Clinical Study to Evaluate the Efficacy and Safety of Carbon Ion Radiotherapy With Atezolizumab and Bevacizumab Combination Therapy in Patients With Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-0048
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Liver Neoplasms; Carcinoma; Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Carcinoma

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-group, open-label, prospective phase II trial evaluating the combination of carbon ion radiotherapy with atezolizumab plus bevacizumab for advanced hepatocellular carcinoma.
Masking Description: This is an open-label study; no masking will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon Ion Radiotherapy + Atezolizumab + Bevacizumab (Experimental): Participants will receive standard first-line systemic therapy with atezolizumab (1200 mg IV every 3 weeks) plus bevacizumab (15 mg/kg IV every 3 weeks). Carbon ion radiotherapy will be integrated as a sequential local treatment during the early phase of systemic therapy.
  Carbon ion radiotherapy will be delivered to the primary hepatic tumor using a hypofractionated regimen (approximately 4-12 fractions), with dose and fractionation individualized according to tumor extent, anatomical proximity to gastrointestinal organs, and institutional organ-at-risk constraints.
  Following completion of carbon ion radiotherapy, participants will continue atezolizumab-bevacizumab maintenance therapy until radiologic disease progression, unacceptable toxicity, or withdrawal of consent. This protocol is designed to enhance local tumor control while preserving the systemic therapeutic benefit of atezolizumab and bevacizumab.
  Interventions: Radiation: Carbon Ion Radiotherapy Atezolizumab Bevacizumab

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy Atezolizumab Bevacizumab — Participants will initiate systemic therapy with atezolizumab (1200 mg IV every 3 weeks) and bevacizumab (15 mg/kg IV every 3 weeks). Carbon ion radiotherapy will subsequently be administered to the primary hepatic lesion during the early phase of systemic therapy.
  Carbon ion radiotherapy will be delivered using a hypofractionated schedule (approximately 4-12 fractions), with dose and fractionation individualized based on tumor size, anatomical location, and organ-at-risk considerations. After completion of carbon ion radiotherapy, participants will continue maintenance treatment with atezolizumab and bevacizumab until disease progression or unacceptable toxicity.
  Other Names: Atezolizumab: Anti-PD-L1 antibody Bevacizumab: Anti-VEGF monoclonal antibody Carbon Ion Radiotherapy: Heavy-ion radiotherapy, C-ion RT

SUMMARY:
This single-center, prospective phase II clinical trial evaluates the safety and therapeutic efficacy of combining carbon ion radiotherapy with the standard first-line regimen of atezolizumab and bevacizumab in patients with advanced hepatocellular carcinoma. The study aims to determine whether the addition of carbon ion radiotherapy enhances tumor control and improves clinical outcomes beyond those achieved with systemic therapy alone. Key endpoints include overall survival, progression-free survival, objective response rate, and treatment-related adverse events.

DETAILED DESCRIPTION:
This clinical trial aims to determine whether adding carbon ion radiotherapy to atezolizumab-bevacizumab therapy improves tumor control and enhances immune response in patients with advanced hepatocellular carcinoma. Over a 3-year study period, eligible patients receiving atezolizumab and bevacizumab who are also suitable for carbon ion radiotherapy will undergo the combined treatment. Clinical outcomes including survival, progression, radiologic response, and toxicity (graded using CTCAE v5.0) will be monitored and assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years Histologically or radiologically confirmed hepatocellular carcinoma (HCC) Barcelona Clinic Liver Cancer (BCLC) stage B or C, not eligible for curative surgery or transplantation.

At least one measurable lesion according to RECIST criteria. Eligible for treatment with atezolizumab plus bevacizumab based on clinical judgment.

Candidate for carbon ion radiotherapy determined by radiation oncologist. Child-Pugh class A liver function Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Adequate organ and marrow function, including:

Absolute neutrophil count ≥ 1,500/μL Platelet count ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min AST/ALT ≤ 5 × ULN Total bilirubin ≤ 3 mg/dL No uncontrolled esophageal or gastric varices, confirmed by endoscopy (within 6 months), or adequately treated before enrollment.

Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

* Prior systemic therapy with anti-PD-1, anti-PD-L1, or anti-VEGF agents within the past year.

Prior carbon ion radiotherapy to the same anatomical region.

Presence of uncontrolled or severe cardiovascular disease, including:

Recent myocardial infarction (within 6 months) Uncontrolled hypertension NYHA class III-IV heart failure Active or history of autoimmune disease requiring systemic immunosuppressive therapy.

Active infection, including:

Uncontrolled bacterial, viral, or fungal infection Active tuberculosis HIV infection, or active hepatitis B/C with uncontrolled viral replication.

Significant bleeding risk, including:

Active gastrointestinal bleeding Untreated or high-risk varices Coagulopathy not controllable with standard therapy Portal vein tumor thrombosis (PVTT) of grade Vp4 if judged unsuitable for treatment by investigator.

Pregnant or breastfeeding women History of organ transplantation, including liver transplantation. Any condition judged by the investigator to interfere with study participation, treatment compliance, or safety evaluation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Three years
  Progression-free survival is defined as the time from the first administration of atezolizumab plus bevacizumab to the date of documented tumor progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | Three years
  Overall survival is defined as the time from the first administration of atezolizumab plus bevacizumab to death from any cause.
  Surviving patients will be censored at the date of the last follow-up. OS defines death or last follow-up date from the date of first AtezoBev administration.
intrahepatic tumor response | Three years
  Tumor response will be evaluated according to RECIST criteria at predefined time points.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): ≥30% decrease in the sum of the longest diameters of target lesions Progressive Disease (PD): ≥20% increase in the sum of the longest diameters of target lesions, or appearance of new lesions Stable Disease (SD): Does not meet criteria for CR, PR, or PD Disease Control Rate (DCR) will be measured as CR + PR + SD. (ORR = CR + PR / DCR = CR + PR + SD)
rate of achieving curative down-staging | Three years
  The proportion of patients who become eligible for curative-intent treatments after tumor down-staging will be assessed.
  Curative treatments may include liver transplantation, hepatic resection, ablation, TACE, or TARE, based on the discretion of the treating physician. How often radical treatments become possible after down-staging A decrease in stage was confirmed during the course of treatment, and treatment targeting the root, such as liver transplantation, hepatic resection, other local ablation, TACE, or TARE, is allowed at the discretion of the physician.
treatment-related toxicity | Three years
  Treatment-related adverse events will be evaluated and graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).
  Safety follow-up will continue from study entry until 30 days after the final planned dose of protocol treatment, or until initiation of subsequent alternative therapy, whichever occurs first.Toxicity is assessed using the National Cancer Society's Common Criteria for Judgment (NCI-CTC). Patients participating in the treatment are subject to safety and toxicity follow-up from participation in the study to 30 days after the final dose of the treatment under the plan is completed (or until the earliest of the start of the next alternative treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No